CLINICAL TRIAL: NCT05627154
Title: Effects of a 14-day Combined Antidepressant and Behavioural Intervention on Emotional Cognition in Healthy Volunteers Experiencing Low Mood
Brief Title: Combined Antidepressant and Behavioural Intervention
Acronym: CABIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: Cabin
Record Dates: First submitted 2022-05-31; First posted 2022-11-25 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Low Mood; Depression; Anxiety
MeSH Terms: conditions — Consciousness Disorders; Depression; Anxiety Disorders | interventions — Citalopram

STUDY DESIGN:
Intervention Model Description: Participants are randomised into one of three groups, each undergoing two weeks of either: 1) placebo alone, 2) citalopram alone or 3) citalopram and behavioural activation training.
Who Masked: Participant, Outcomes Assessor
Masking Description: Due to the nature of the intervention, the study will be single blinded only to citalopram or placebo administration. As the primary researcher will be the one administering the behavioural activation (BA) training, both the participants and the primary researcher will be aware of who did or did not receive the psychological intervention. However, participants will not be aware that receiving BA means they are also taking citalopram. The primary researcher, on the other hand, will be aware of this and will only be blinded to drug administration in the BA-free groups. To compensate for the lack of complete blinding, post-treatment outcome data will be collected online and not directly by the primary researcher. Moreover, before the data is analysed, participant ID numbers will be re-allocated to avoid bias in the outlier detection and data exclusion process.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Placebo only (Placebo Comparator): Participants randomised to the Placebo condition will be taking a lactose placebo capsule daily for 14 days.
  Interventions: Drug: Placebo
- Citalopram only (Experimental): Participants randomised to the Citalopram only condition will be taking 20mg of citalopram in capsule form daily for 14 days.
  Interventions: Drug: Citalopram
- Citalopram and Behavioural Activation (Experimental): Participants randomised to the Citalopram only condition will be taking 20mg of citalopram in capsule form daily for 14 days. Over the two weeks of taking citalopram, they will also receive ~3h of behavioural activation therapy split into 3 sessions.
  Interventions: Drug: Citalopram; Behavioral: Behavioural Activation

INTERVENTIONS:
Drug: Citalopram — Serotonin-reuptake inhibitor commonly used to treat depressive and anxiety disorders.
  Arms: Citalopram and Behavioural Activation; Citalopram only
Behavioral: Behavioural Activation — A NICE recommended psychological intervention for mild to moderate depression. In behavioural activation, the person with depression and the therapist work together to identify the relationships between the activities the person undertakes and their mood. It encourages people to become less mood-dependent when planning activities and doing constructive things that they would usually avoid doing.
  Arms: Citalopram and Behavioural Activation
Drug: Placebo — A lactose-based tablet.
  Arms: Placebo only

SUMMARY:
A body of evidence from both animal and human research suggests that antidepressant drugs may induce early changes in emotional processing that interact with environmental factors to produce a later change in mood. This experimental medicine study will examine the effect of citalopram on emotional cognition under different environmental conditions (as manipulated by the presence or absence of behavioural activation training). Participants will be administered either citalopram or placebo over the course of two weeks. Citalopram will be taken either alone or in combination with behavioural activation training.

DETAILED DESCRIPTION:
Major Depressive Disorder (MDD) is a common psychiatric condition characterised by pervasive low mood as well as changes in sleep, appetite and cognition. In the UK, it is estimated that 3 in 100 people meet criteria for MDD every week, costing the economy £20.2-23.8 billion every year in health service, lost earnings and lower productivity.

A variety of pharmacological and psychological interventions for MDD are available. Selective serotonin reuptake inhibitors (SSRIs) are the first-choice medication for depression in the UK, as recommended by National Institute of Health and Care Excellence (NICE) guidelines. Whilst SSRIs have been demonstrated to be more effective than placebo, only about 50% of patients respond to their first-prescribed antidepressant. Understanding the mechanism through which SSRIs exert their antidepressant effect could explain why their effectiveness is not universal and allow for personalised treatments.

Experimental medicine studies conducted over the last 15-20 years have shown that SSRIs have early effects on emotional cognition, and that these precede clinically significant changes in depressive symptomatology. For example, one week of treatment with citalopram was found to decrease recognition of negative facial expressions and increase the relative recall of positive vs negative words. The switch from implicit changes in cognitive bias to explicit changes in mood is thought to occur through interaction with the environment and re-learning of positive associations. Indeed, rodent studies suggest that SSRIs only induce a positive bias in memory when administered before learning and that SSRI-induced neuroplasticity only occurs in the presence of an positive/enriched environment.

These findings imply that an enriched environment from which patients can derive positive and meaningful reinforcement may be important for antidepressant function. This hypothesis is indirectly supported by multiple reports of a positive correlation between antidepressant treatment outcome and patients' socioeconomic status as a proxy for environmental enrichment, but to our knowledge this has not been experimentally tested in humans.

This experimental medicine study will explore whether the early cognitive effects of the SSRI citalopram are modulated by different levels of environmental enrichment. The presence/absence of environmental enrichment will be modulated through provision of two weeks of behavioural activation (BA) training to a third of our sample; BA is a psychological intervention aimed to increase levels of environmental reinforcement by monitoring and adjusting an individual's daily activities. By comparing the combined effects of citalopram and BA to those of citalopram alone and placebo alone on performance of emotional cognition tasks (Emotional Test Battery (ETB)), the investigators will test whether the early cognitive changes induced by antidepressants are increased in the context of a more rewarding environment. The investigators hypothesise that the participant group receiving citalopram and BA will show greater changes in emotional cognition in the expected direction (decrease in negative bias/increase in positive bias) compared to the citalopram alone and placebo alone groups after the two-week intervention.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-65 years inclusive
* Resident in the UK for the duration of the study
* Fluent in English
* Normal or corrected-to-normal vision
* Experiencing subjective low mood (score of 10 or above on the BDI-II)
* Experiencing low activity levels (self-reported)
* Willing and able to give informed consent for participation in the research
* Access to a computer or laptop with a functioning keyboard and a reliable internet connection

Exclusion Criteria:

* Antidepressant treatment or medication prescribed to treat depression/low mood, currently or in the last six months
* Current psychological therapy of any kind
* Current or past probable diagnosis of psychosis, bipolar disorder, OCD, PTSD, substance abuse disorder or any eating disorder, as indicated by the SCID-5
* Current or past diagnosis of any personality disorder (e.g. borderline personality disorder) according to self-report
* Judged to be at clinical high risk of suicide
* Past suicide attempt
* Current or past hospitalisation for mental health reasons
* 1st degree relative with diagnosis of bipolar disorder
* Diagnosis of a developmental disorder (e.g. ASD, ADHD, Tourette's syndrome, severe learning disability) according to self-report; this excludes cases of mild dyslexia or dyscalculia where in the opinion of the study team such difficulties would not interfere with the performance of the tasks required in this study
* Diagnosis of a neurological disorder (e.g. epilepsy, MS) according to self-report
* Score of >30 on the BDI-II
* Current use of medication that might interact with the effects of citalopram (except for the contraceptive pill)
* Known contraindication to citalopram including: past allergic reaction to citalopram or any other medicines, diagnosis of a cardiovascular condition, glaucoma, type 1 or type 2 diabetes, diagnosis of epilepsy, undergoing electroconvulsive treatment (ECT), or current use of any other medication that is associated with prolonged QT-interval
* Any other current or past medical conditions which in the opinion of the study medic may interfere with the safety of the participant or the scientific integrity of the study
* Heavy use of cigarettes (smoke > 20 cigarettes per day)
* Heavy use of caffeine (drink > 4 250ml cups/cans of coffee/energy drinks per day)
* Severely underweight or overweight in a manner that renders them unsuitable for the study in the opinion of the study medic
* Lactose intolerance (due to the study involving administration of a lactose placebo tablet)
* Pregnancy (as determined by urine pregnancy test taken during the Part 2 screening visit), breast feeding or plans to become pregnant
* Participation in an ETB study in the past 6 months
* Participation in another drug study in the past 3 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2021-05-28 (Actual); Primary Completion 2023-11-17 (Actual); Study Completion 2023-11-17 (Actual)

PRIMARY OUTCOMES:
Changes in emotional cognition | Pre-intervention and 13-15 days after the start of the intervention
  Accuracy and reaction times on computer-based measures of emotional cognition (facial expression recognition task, emotional word categorisation task, emotional word recall task, emotional word recognition task).

SECONDARY OUTCOMES:
Changes in reward processing | Pre-intervention and 13-15 days after the start of the intervention
  Accuracy, consistency, reaction times, monetary wins and losses, learning rate and decision temperature on the Probabilistic Instrumental Learning Task.
Changes in motor activity | 7 days pre-intervention compared to last 7 days of intervention
  Acceleration, light and temperature data measured at 25 Hz using GENEActiv actigraphy watches
Changes in salivary cortisol | Pre-intervention and 13-14 days after the start of the intervention
  Waking cortisol levels assayed using a Salimetrics Salivary Cortisol ELISA Kit from 6 saliva samples (3 pre- and 3 post-intervention) collected using Sarstedt Salivette® Cortisol tubes

OTHER OUTCOMES:
Changes in daily mood | 7 days pre-intervention compared to last 7 days of intervention
  Fluctuations in daily mood measures using a Mood Zoom format, comprising six items on a 7-point Likert scale

CONTACTS AND LOCATIONS:
Overall Officials: Catherine J Harmer, DPhil, Principal Investigator — Department of Psychiatry, University of Oxford
Locations (1):
- Neurosciences Building, Warneford Hospital, Oxford, Oxfordshire, United Kingdom

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-03-31): https://cdn.clinicaltrials.gov/large-docs/54/NCT05627154/Prot_SAP_000.pdf
  • Informed Consent Form (2021-03-23): https://cdn.clinicaltrials.gov/large-docs/54/NCT05627154/ICF_001.pdf